CLINICAL TRIAL: NCT01323881
Title: Theta Burst Stimulation on the Motor Cortex in Acute Stroke: a Randomized Controlled Trial
Brief Title: Intermittent Theta Burst Stimulation After Acute Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, I-Hui Lee, MD PhD, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGHIRB98-05-05
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2009-05

CONDITIONS: Ischemic Stroke,
Keywords: theta burst stimulation, stroke, motor, plasticity
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intermittent theta burst stimulation (Experimental)
  Interventions: Device: Intermittent theta burst stimulation
- sham stimulation (Placebo Comparator)

INTERVENTIONS:
Device: Intermittent theta burst stimulation — Intermittent theta burst stimulation with 1200 pulses or sham stimulation over the ipsilesional M1 hand region for 10 daily sessions in 2 weeks.
  Arms: intermittent theta burst stimulation

SUMMARY:
This pilot sham-controlled study aims to determine the safety and efficacy of repetitive transcranial magnetic stimulation given as a facilitatory intermittent theta burst stimulation (iTBS1200, 1200 stimuli/session) paradigm to enhance motor recovery in subacute stroke patients.

DETAILED DESCRIPTION:
The patients with first-ever, MRI-confirmed monohemispheric ischemic stroke in the middle cerebral artery territory, and NIH Stroke Scale motor arm score 1-2 with recordable active motor thresholds (aMT) of the extensor carpi radialis (ECR) between 2-4 weeks after the stroke onset, are randomized into two groups to receive either iTBS1200 or sham stimulation over the ipsilesional M1 hand region for 10 daily sessions in 2 weeks. All have standardized medical and intensive rehabilitation treatments. The outcome measures included Action Research Arm test (ARAT), Fugl-Meyer test (FMT), aMT and motor evoked potentials (MEPs) of ECR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first-ever, subacute (between 2-4 weeks post-stroke), monohemispheric ischemic stroke within the middle cerebral artery (MCA) territory, and mild to moderate hand paresis (NIHSS motor arm score 1-2) are enrolled.

Exclusion Criteria:

* age over 75, severe hand paresis without detectable active motor threshold (aMT) of the extensor carpi radialis (ECR), seizure history (clinical or EEG abnormalities), psychosis, aphasia, apraxia, concomitant neurological diseases or severe systemic diseases (e.g. sepsis, advanced malignancy, hepatic or renal failure.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The changes of Action Research Arm test | 60th day post-stroke
  We assess the changes of Action Research Arm test between before the intervention and the 60th day post-stroke.

SECONDARY OUTCOMES:
The changes of upper limb function and corticospinal excitability | 60th day post-stroke
  We assess the changes of Fugl-Meyer test (FMT), active motor threshold and motor evoked potentials (MEPs) of paretic ECR between before the intervention and 60th day post-stroke

CONTACTS AND LOCATIONS:
Overall Officials: I-Hui Lee, MD PhD, Principal Investigator — Department of Neurology, Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Hsu YF, Huang YZ, Lin YY, Tang CW, Liao KK, Lee PL, Tsai YA, Cheng HL, Cheng H, Chern CM, Lee IH. Intermittent theta burst stimulation over ipsilesional primary motor cortex of subacute ischemic stroke patients: a pilot study. Brain Stimul. 2013 Mar;6(2):166-74. doi: 10.1016/j.brs.2012.04.007. Epub 2012 May 12. PMID 22659021